CLINICAL TRIAL: NCT01079455
Title: Comparison of Hyaluronic Acid and Corticosteroid Intra-articular Injections for the Treatment of Osteoarthritis of the Hip Controlled With Intra-articular Injections With Bupivacaine
Brief Title: Comparison of Hyaluronic Acid and Corticosteroid Intra-articular Injections for the Treatment of Osteoarthritis of the Hip
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Pellenberg (Other)
Responsible Party: University Hospital Pellenberg, University Hospital Pellenberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-014274-17
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-02

CONDITIONS: Coxarthrosis
Keywords: Coxarthrosis; Hip; Infiltration; Hyaluronic Acid; Corticosterone
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Corticosterone; Hyaluronic Acid; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HA (Active Comparator): Coxarthrosis
  Interventions: Drug: Corticosterone
- Corticosterone (Active Comparator): Coxarthrosis
  Interventions: Drug: Corticosterone
- Bupivacaine (Placebo Comparator): Coxarthrosis
  Interventions: Drug: Corticosterone

INTERVENTIONS:
Drug: Corticosterone — Hyaluronic acid 40 mg / 2 ml Corticosteroids 80 mg / 2 ml Bupivacaine 0.125% / 2 ml
  Other Names: Hyaluronic Acid; Bupivacaine

SUMMARY:
Abstract Background: The effect of intra-articular treatment of hip osteoarthritis with hyaluronic acid in the hip joint is not based on large randomized controlled trials. Hyaluronic acid is a well established treatment for osteoarthritis of the knee.

Methods: Randomized controlled trial with three-armed parallel-group design. The patients meeting the inclusion criteria will be randomized into one of the following groups: infiltration of the hip joint with hyaluronic acid, with corticosteroids or with bupivacaine 0,125%.

Pain VAS, Harris Hip Score and HOOS were scored during follow-up. The patients will be asked to determine their situation as worse, stabile or better then at the time of enrollment. There will be asked if they use painkillers and if they have complications/adverse events. These outcome measure instruments will be used at the time of enrollment in the study prior to any injection, and then again at six weeks, 3 and 6 months after the initial injection. The six-month follow-up period begins for all patients on the date the first injection will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. an age between 30 and 70years
2. radiographic evidence of OA of the hip (Kellgren-Lawrence grading scale 1-3)
3. chronic pain for at least 3 months prior to study entry (day 0)
4. dissatisfaction with prior attempts at non-operative management including nonsteroidal anti-inflammatory drugs.

Exclusion Criteria:

1. Kellgren and Lawrence grade 4
2. an intra-articular hip injection (with any corticosteroid, hyaluronic acid preparation or other) within the previous three months
3. non compliance to the study procedures and or non completion of the study according to investigator's judgment
4. rapid destructive hip.
5. a history of crystalline arthropathy or inflammatory arthritis, neuropathic arthropathy
6. a current other problem in the affected extremity
7. contra-indications for the use of corticosteroids (gastrointestinal ulcer, severe osteoporosis, psychiatric anamnesis, herpes simplex or zoster (viremic stadium), varicella, 8 weeks before and 2 weeks after immunization, systemic mycosis, poliomyelitic except of bulbar encephalitic form lymphadenitis after BCG-vaccination, parenteral depot medication, closed- and wide-angle glaucoma)
8. allergy or hypersensitivity to any of the study medications or to contrast solutions.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 0 - 6 - 12 - 26 weeks
  this score will be used as a self-administered questionnaire in accordance with the developers' instructions. The Harris Hip Score was first developed in 1967 and is accepted as one of the best used questionnaires dealing the hip function. It is a disease-specific scoring system which was introduced to provide an evaluation system for various hip disabilities and methods of treatment. This Score gives a maximum of 100 points, with domains of pain, function, deformity and motion.

SECONDARY OUTCOMES:
Visual Analog Score | 0 - 6 - 12 - 26 weeks
  this score is a self-assessment of variation in pain intensity, measured on a simple 100-mm-long continuous scale of absolutes ranging from "no pain" to "extreme pain". The percentage of pain is determined by physical measuring from the end of the line to the patients' mark on the pain scale, and divided by total length of the line. The advantage of the VAS is that you can determine the change in pain by taking the difference between any two recordings of pain severity

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Colen, MD, Principal Investigator — University Hospital Pellenberg
Locations (1):
- University Hospital Pellenberg, Leuven, Belgium

REFERENCES:
- [Derived] Colen S, van den Bekerom MP, Bellemans J, Mulier M. Comparison of intra-articular injections of hyaluronic acid and corticosteroid in the treatment of osteoarthritis of the hip in comparison with intra-articular injections of bupivacaine. Design of a prospective, randomized, controlled study with blinding of the patients and outcome assessors. BMC Musculoskelet Disord. 2010 Nov 16;11:264. doi: 10.1186/1471-2474-11-264. PMID 21080920